CLINICAL TRIAL: NCT02985723
Title: Prospective Study to Evaluate the Visual Outcome, Cylinder Correction and Patient Satisfaction After Implantation of AT LISA Tri Toric 939MP Intraocular Lenses
Brief Title: Visual Outcome, Cylinder Correction and Patient Satisfaction After Implantation of AT LISA Tri Toric 939MP Intraocular Lenses
Acronym: VICTORI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-A01671-42
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

ARMS (1):
- 939MP (Experimental): AT LISA tri toric 939MP intraocular lens
  Interventions: Device: AT LISA tri toric 939MP

INTERVENTIONS:
Device: AT LISA tri toric 939MP

SUMMARY:
The aim of the present study is to evaluate the postoperative visual acuity for distance, intermediate and near vision as well as the cylinder correction and the patient satisfaction after bilateral implantation of AT LISA tri toric 939MP IOLs.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed of the consequences and constraints of the protocol and who has given his/her written informed consent
* Man or woman, over 50 years of age
* Healthy eyes with bilateral cataract requiring surgical treatment for both eyes
* Bilateral regular corneal astigmatism (confirmed by topography measurement)
* Only patients requiring intraocular lenses of a power comprised between sphere +0.0 and +28.0 dioptres and between a cylindrical range of +1.0 to +4.0D in both eyes will be able to participate in the trial.
* Biometry measurement/cataract density compatible with the IOLMaster evaluation
* Bilateral uncomplicated cataract surgery and implantation into capsular bag by injector
* Assured follow-up examinations

Exclusion Criteria:

* Patients unable to meet the limitations of the protocol or likely of non cooperation during the trial,
* Patients whose freedom is impaired by administrative or legal order,
* Monophtalmic patient.
* Previous ocular surgery, including corneal/refractive surgery,
* Chronic or recurrent uveitis,
* Acute ocular disease or external/internal infection,
* Any kind of macular degeneration and impairment of retina (clinical diagnosis/OCT examination)
* Diabetes with retinal changes,
* Pseudoexfoliation syndrome
* Pathologic myosis
* Irregular astigmatism, especially keratoconus,
* Endothelial corneal dystrophy
* Glaucoma or IOP higher than 21mmHg under ocular hypertension treatment
* Aniridia
* Pseudophakia
* Cornea guttata; keratoplasty
* Amotio operation; anamnesis with vitreous surgery
* Amblyopia
* Intraocular tumours; endotamponade
* Phlogistic intraocular processes or other pre-existing processes that permanently limit the best corrected visual acuity to > 0.3 logMAR
* Any other pathology or condition presenting, according to the investigator opinion, a risk for the patient
* Pupil diameter over 6 mm in mesopic condition
* Corneal opacity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Best distance-corrected visual acuity for intermediate vision after bilateral implantation | 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Piovella, Dr, Principal Investigator — CMA - Centro Microchirurgia Ambulatoriale